CLINICAL TRIAL: NCT02032277
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase 3 Study Evaluating Safety and Efficacy of the Addition of Veliparib Plus Carboplatin Versus the Addition of Carboplatin to Standard Neoadjuvant Chemotherapy Versus Standard Neoadjuvant Chemotherapy in Subjects With Early Stage Triple Negative Breast Cancer (TNBC)
Brief Title: A Study Evaluating Safety and Efficacy of the Addition of ABT-888 Plus Carboplatin Versus the Addition of Carboplatin to Standard Chemotherapy Versus Standard Chemotherapy in Subjects With Early Stage Triple Negative Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: GBG Forschungs GmbH (Other); NSABP Foundation Inc (Network); Grupo Español de Investigación del Cáncer de Mama (Unknown); US Oncology Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-011; 2013-002377-21 (EudraCT Number)
Expanded Access: NCT03123211 (No longer available)
Record Dates: First submitted 2013-12-13; First posted 2014-01-10 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Triple Negative Breast Cancer
Keywords: Oncology; Triple negative breast cancer; German Breast Group - GBG 81; United States Oncology - 12152; National Surgical Adjuvant Breast and Bowel Project - B-56-I; Alliance - AFT-04; Grupo Español de Investigación en Cáncer de Mama - GEICAM/2014-02
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Paclitaxel; Carboplatin; veliparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A (Active Comparator): Veliparib + carboplatin + paclitaxel followed by doxorubicin/cyclophosphamide (AC)
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Paclitaxel; Drug: Carboplatin; Drug: Veliparib
- Arm C (Placebo Comparator): Placebo + placebo + paclitaxel followed by AC.
  Interventions: Drug: Cyclophosphamide; Drug: Placebo; Drug: Doxorubicin; Drug: Paclitaxel
- Arm B (Placebo Comparator): Placebo + carboplatin + paclitaxel followed by AC
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Paclitaxel; Drug: Carboplatin; Drug: Placebo

INTERVENTIONS:
Drug: Cyclophosphamide — Cyclophosphamide
Drug: Placebo — Placebo for Carboplatin
  Arms: Arm C
Drug: Doxorubicin — Doxorubicin
Drug: Paclitaxel — Paclitaxel
Drug: Carboplatin — Carboplatin
  Arms: Arm A; Arm B
Drug: Veliparib — Veliparib
  Other Names: ABT-888
  Arms: Arm A
Drug: Placebo — Placebo for Veliparib
  Arms: Arm B; Arm C

SUMMARY:
This is a 3 arm Phase 3 study to evaluate the safety and efficacy of the addition of veliparib plus carboplatin versus the addition of carboplatin to standard neoadjuvant chemotherapy versus standard neoadjuvant chemotherapy in subjects with early stage TNBC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer by core needle or incisional biopsy (excisional biopsy is not allowed). Clinical stage T2-3 N0-2 or T1 N1-2 by physical exam or radiologic studies.
2. Documented Breast Cancer Gene (BRCA) germline mutation testing.
3. Estrogen Receptor (ER)-, Progesterone Receptor (PR)-, and Human Epidermal Growth Factor Receptor (HER)2-negative (triple-negative) cancer of the breast.
4. ECOG Performance status of 0 to 1.
5. Women must be determined to be not of childbearing potential (surgically sterile, or postmenopausal defined as amenorrheic for at least 12 months) by the Investigator OR they must have a negative serum pregnancy test prior to randomization.

Exclusion Criteria:

1. Previous anti-cancer treatment (cytotoxic chemotherapy, immunotherapy, biologic therapy radiotherapy or investigational agents) with therapeutic intent for current breast cancer.
2. Previous treatment with carboplatin, paclitaxel, doxorubicin, cyclophosphamide and a Poly-(ADP-ribose)-Polymerase (PARP) inhibitor.
3. Concurrent treatment with an ovarian hormonal replacement therapy or with hormonal agents such as raloxifene, tamoxifen or other selective estrogen receptor modulator (SERM). Subjects must have discontinued use of such agents prior to beginning study treatment.
4. A history of seizure within 12 months prior to study entry.
5. Pre-existing neuropathy from any cause in excess of Grade 1.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2016-03-18 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR). | At the time of definitive surgery (approximately 24-36 weeks from first dose of study drug).
  Pathological complete response (pCR) in the breast tissue and the lymph node tissue will be assessed upon completion of pre-operative systemic therapy and definitive surgery.

SECONDARY OUTCOMES:
Event Free Survival (EFS) | Up to 4 years from the date of definitive surgery.
  EFS will be defined as the time from random assignment to documentation of the first of the following events: discontinuation of study therapy due to protocol-defined progression prior to surgery; local, regional, or distant recurrence of breast cancer following curative surgery; a new breast cancer; another new onset malignancy; or death as a result of any cause.
Overall Survival (OS) | Up to 4 years from the date of definitive surgery.
  OS will be defined as the number of days from the day the subject is randomized to the date of the subject's death.
Rate of eligibility for breast conservation after therapy (BCR). | At the time of definitive surgery (approximately 24-36 weeks from first dose of study drug).
  Whether a subject is eligible for breast conserving surgery for whom mastectomy was planned at diagnosis will be determined by the subject's surgeon prior to chemotherapy and after completion of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (158):
- United States (61):
  - Scottsdale Healthcare /ID# 120473, Scottsdale, Arizona
  - Mayo Clinic - Scottsdale /ID# 139932, Scottsdale, Arizona
  - Arizona Oncology Associates, PC-HOPE /ID# 126137, Tucson, Arizona
  - Usc /Id# 123310, Los Angeles, California
  - Pacific Cancer Care /ID# 120476, Salinas, California
  - Sharp Memorial Hospital /ID# 119861, San Diego, California
  - Stanford University School of Med /ID# 130316, Stanford, California
  - Cedars-Sinai Medical Center - West Hollywood /ID# 137275, West Hollywood, California
  - Christiana Care Health Service /ID# 137823, Newark, Delaware
  - Florida Cancer Specialists - Fort Myers /ID# 121835, Fort Myers, Florida
  - Florida Cancer Specialists - Fort Myers /ID# 126379, Fort Myers, Florida
  - Mayo Clinic /ID# 132349, Jacksonville, Florida
  - Mount Sinai Comp Cancer Ctr /ID# 133008, Miami, Florida
  - Miami Cancer Institute - Baptist Health South Florida /ID# 126145, Miami, Florida
  - UF Health Cancer Center /ID# 141589, Orlando, Florida
  - Moffitt Cancer Center /ID# 124063, Tampa, Florida
  - University of Illinois - Chicago /ID# 134329, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 133848, Chicago, Illinois
  - University of Chicago DCAM /ID# 120467, Chicago, Illinois
  - Loyola University Medical Ctr /ID# 120455, Maywood, Illinois
  - OSF St. Anthony Medical Center /ID# 139424, Rockford, Illinois
  - Indiana Univ School Medicine /ID# 118215, Indianapolis, Indiana
  - Community Rgnal Cancer Care N /ID# 120456, Indianapolis, Indiana
  - Horizon Oncology Research Center /ID# 116815, Lafayette, Indiana
  - Cancer Center of Kansas /ID# 134720, Wichita, Kansas
  - Univ Maryland School Medicine /ID# 119235, Baltimore, Maryland
  - St. Joseph Mercy Hospital /ID# 135875, Ypsilanti, Michigan
  - Minnesota Oncology Hematology, PA /ID# 126144, Minneapolis, Minnesota
  - St. Lukes Cancer Institute /ID# 118775, Kansas City, Missouri
  - Comprehensive Cancer Ctrs Neva /ID# 126136, Las Vegas, Nevada
  - Solinksy Center for Cancer Care /ID# 131970, Manchester, New Hampshire
  - Rutgers Cancer Institute of NJ /ID# 120477, New Brunswick, New Jersey
  - Columbia Univ Medical Center /ID# 141588, New York, New York
  - Hope Womens Cancer Centers /ID# 119179, Asheville, North Carolina
  - Univ NC Chapel Hill /ID# 132893, Chapel Hill, North Carolina
  - Univ NC Chapel Hill /ID# 147695, Chapel Hill, North Carolina
  - Novant Health Oncology Special /ID# 139890, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Cen /ID# 132394, Fargo, North Dakota
  - Oncology Hematology Care, Inc - Blue Ash /ID# 120478, Cincinnati, Ohio
  - University Hospitals Case Medical Center /ID# 141691, Cleveland, Ohio
  - Fairview Hospital /ID# 141626, Cleveland, Ohio
  - Cleveland Clinic Main Campus /ID# 126378, Cleveland, Ohio
  - The Ohio State University /ID# 141587, Columbus, Ohio
  - Lehigh Valley Health Network /ID# 133372, Allentown, Pennsylvania
  - Guthrie Medical Group, PC /ID# 124397, Sayre, Pennsylvania
  - Women and Infants Hospital /ID# 123476, Providence, Rhode Island
  - Avera Cancer Institute /ID# 120466, Sioux Falls, South Dakota
  - Tennessee Oncology, PLLC /ID# 124566, Nashville, Tennessee
  - Texas Oncology - Bedford /ID# 126135, Bedford, Texas
  - Texas Oncology - Medical City Dallas /ID# 126140, Dallas, Texas
  - Texas Oncology - Medical City Dallas /ID# 126141, Dallas, Texas
  - UT Southwestern Medical Center /ID# 133849, Dallas, Texas
  - The Ctr for Cancer and Blood D /ID# 120479, Fort Worth, Texas
  - Texas Oncology - Memorial City /ID# 126139, Houston, Texas
  - Texas Oncology - Plano East /ID# 126143, Plano, Texas
  - Texas Oncology - Tyler /ID# 126142, Tyler, Texas
  - University of Utah /ID# 118677, Salt Lake City, Utah
  - University of Virginia /ID# 122975, Charlottesville, Virginia
  - Virginia Commonwealth Univ /ID# 141586, Richmond, Virginia
  - Virginia Oncology Associates /ID# 127260, Virginia Beach, Virginia
  - Univ of Wisconsin Hosp/Clinics /ID# 120457, Madison, Wisconsin
- Australia (7):
  - The Tweed Hospital /ID# 120235, Tweed Heads, New South Wales
  - Cabrini Health /ID# 120236, Malvern, Victoria
  - Royal Melbourne Hospital /ID# 127717, Parkville, Victoria
  - Western Health Sunshine Hosp. /ID# 120715, St Albans, Victoria
  - Fiona Stanley Hospital /ID# 120716, Murdoch, Western Australia
  - St. John of God Hosp - Murdoch /ID# 131788, Murdoch, Western Australia
  - St. John of God Subiaco Hosp /ID# 120717, Subiaco, Western Australia
- Belgium (6):
  - Cliniques Universitaires Saint Luc /ID# 120719, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hôpital de Charleroi /ID# 116678, Charleroi, Hainaut
  - CHU Brugmann /ID# 120376, Brussels
  - UZ Antwerp /ID# 120720, Edegem
  - AZ Groeninge /ID# 120718, Kortrijk
  - CHU UCL Namur /ID# 116677, Namur
- Canada (4):
  - Sunnybrook Health Sciences Ctr /ID# 123312, Toronto, Ontario
  - CHUM - Notre-Dame Hospital /ID# 141694, Montreal, Quebec
  - Jewish General Hospital /ID# 141629, Montreal, Quebec
  - CHUQ-Hospital St. Sacrement /ID# 141619, Québec, Quebec
- Czechia (3):
  - Fakultni Nemocnice Olomouc /ID# 120725, Olomouc, Olomoucký kraj
  - Masarykuv onkologikcy ustav /ID# 120726, Brno
  - FN Hradec Kralove /ID# 120596, Hradec Králové
- France (7):
  - Hopital Universitaire Purpan /ID# 120731, Toulouse, Haute-Garonne
  - Centre Oscar Lambret /ID# 119958, Lille, Hauts-de-France
  - Centre Leon Berard /ID# 120740, Lyon, Rhone
  - Jean Perrin Centre /ID# 125277, Clermont-Ferrand
  - Hosp European, Georges Pompid /ID# 120736, Paris
  - Hopital Rene Huguenin /ID# 120729, Saint-Cloud
  - Institut Curie /ID# 116679, Paris, Île-de-France Region
- Germany (20):
  - Universitaetsklinikum Schleswig-Holstein /ID# 133454, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Ulm /ID# 133453, Ulm, Thuringia
  - Gemeinschaftspraxis Dr. Heinrich und Prof. Bangerter /ID# 133472, Augsburg
  - Helios Klinikum Berlin Buch /ID# 133465, Berlin
  - Studiengesellschaft Onk Bielef /ID# 133471, Bielefeld
  - Klinikum Bremen Mitte gGmbH /ID# 132875, Bremen
  - St. Johannes Hospital /ID# 133478, Dortmund
  - Kliniken Esslingen /ID# 133475, Esslingen am Neckar
  - Klinikum Frankfurt Hoechst /ID# 145301, Frankfurt
  - Wilke/Wagner/Petzoldt, Fuerth /ID# 133481, Fürth
  - Evangelisches Krankenhaus /ID# 133457, Gelsenkirchen
  - Elisabeth Krankenhaus /ID# 133461, Kassel
  - St. Vincenz Krankenhaus /ID# 133466, Limburg
  - Onk Zentrum am Rotkreuz /ID# 133482, Munich
  - Klinikum recht der Isar der TU /ID# 133449, Munich
  - Sana Klinikum Offenbach /ID# 133455, Offenbach
  - Leopoldina-Krankenhaus /ID# 133484, Schweinfurt
  - Johanniter-Krankenhaus Genthin /ID# 133463, Stendal
  - St. Josefs-Hospital /ID# 133464, Wiesbaden
  - Marienhospital Witten /ID# 133470, Witten
- Hungary (9):
  - National Institute of Oncology /ID# 120828, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont /ID# 120834, Budapest
  - Uzsoki Utcai Korhaz /ID# 120825, Budapest
  - Debreceni Egyetem Klinikai Kozpont /ID# 116681, Debrecen
  - Petz Aladar Megyei Oktato Korh /ID# 120835, Győr
  - Bacs-Kiskun Megyei Korhaz /ID# 120833, Kecskemét
  - BAZ Megyei E.O. Korhaz /ID# 122215, Miskolc
  - University of Szeged /ID# 120823, Szeged
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz /ID# 120818, Szolnok
- Italy (5):
  - A.O.U. Policlinico S.Orsola-Malpighi /ID# 122855, Bologna, Emilia-Romagna
  - Misericordia General Hospital /ID# 119536, Grosseto
  - IRCCS-I.R.S.T. srl Meldola /ID# 120255, Meldola
  - Istituto Europeo di Oncologia /ID# 120845, Milan
  - IRCCS Fondazione Salva Maugeri /ID# 120848, Pavia
- Vrije Universiteit Medisch Centrum /ID# 126302, Amsterdam, Netherlands
- Russia (7):
  - Federal State Budgetary Scientific Institution N.N. Blokhin Russian Cancer Resea /ID# 120944, Moscow, Moscow
  - Kursk Regional Oncology Dispen /ID# 116688, Kursk, Tatarstan, Respublika
  - archangel Clinical Oncology /ID# 120935, Arkhangelsk
  - Medical Radiological Res Ctr /ID# 124017, Obninsk
  - Pyatigorsk Oncology Dispensary /ID# 120945, Pyatigorsk
  - Leningrad Reg Onc Dispensery /ID# 120938, Saint Petersburg
  - Birch A Healthcare /ID# 116695, Saint Petersburg
- South Korea (8):
  - National Cancer Center /ID# 119525, Goyang, Gyeonggido
  - Ajou University Hospital /ID# 118856, Suwon, Gyeonggido
  - Kyungpook National University Chilgok Hospital /ID# 118855, Daegu, Seoul Teugbyeolsi
  - Severance Hospital /ID# 116699, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 119276, Seoul, Seoul Teugbyeolsi
  - Korea University Anam Hospital /ID# 118857, Seoul
  - Seoul National University Hospital /ID# 116698, Seoul
  - Asan Medical Center /ID# 116696, Seoul
- Spain (13):
  - Hospital Universitario A Coruña - CHUAC /ID# 135108, A Coruña, A Coruna
  - Hospital Universitario Germans Trias i Pujol /ID# 135112, Badalona, Barcelona
  - Hospital General Universitario Alicante /ID# 135115, Alicante
  - Hospital Parc de Salut del Mar /ID# 135110, Barcelona
  - Hospital Santa Creu i Sant Pau /ID# 145400, Barcelona
  - Hospital Universitario Arnau de Vilanova de Lleida /ID# 120979, Lleida
  - Hospital Universitario Ramon y Cajal /ID# 135113, Madrid
  - Hospital Clinico Universitario San Carlos /ID# 119959, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 135114, Seville
  - Fundacion Instituto Valenciano Oncologia IVO /ID# 135116, Valencia
  - Hospital Clinico Universitario de Valencia /ID# 123076, Valencia
  - Hospital General Universitario de Valencia /ID# 135111, Valencia
  - Hospital Universitario Miguel Servet /ID# 119195, Zaragoza
- Taiwan (3):
  - National Taiwan Univ Hosp /ID# 122895, Taipei City, Taipei
  - Changhua Christian Hospital /ID# 119085, Changhua County
  - Chi Mei Hospital - Liouying /ID# 120982, Tainan
- United Kingdom (4):
  - Univ Hosp Bristol NHS Foundati /ID# 120989, Bristol
  - Charing Cross Hospital /ID# 120990, London
  - Nottingham Univ Hospitals NHS /ID# 122218, Nottingham
  - Royal Stoke Univ Hospital /ID# 120984, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Filho OM, Stover DG, Asad S, Ansell PJ, Watson M, Loibl S, Geyer CE Jr, Bae J, Collier K, Cherian M, O'Shaughnessy J, Untch M, Rugo HS, Huober JB, Golshan M, Sikov WM, von Minckwitz G, Rastogi P, Maag D, Wolmark N, Denkert C, Symmans WF. Association of Immunophenotype With Pathologic Complete Response to Neoadjuvant Chemotherapy for Triple-Negative Breast Cancer: A Secondary Analysis of the BrighTNess Phase 3 Randomized Clinical Trial. JAMA Oncol. 2021 Apr 1;7(4):603-608. doi: 10.1001/jamaoncol.2020.7310. PMID 33599688
- [Derived] Golshan M, Loibl S, Wong SM, Houber JB, O'Shaughnessy J, Rugo HS, Wolmark N, McKee MD, Maag D, Sullivan DM, Metzger-Filho O, Von Minckwitz G, Geyer CE Jr, Sikov WM, Untch M. Breast Conservation After Neoadjuvant Chemotherapy for Triple-Negative Breast Cancer: Surgical Results From the BrighTNess Randomized Clinical Trial. JAMA Surg. 2020 Mar 1;155(3):e195410. doi: 10.1001/jamasurg.2019.5410. Epub 2020 Mar 18. PMID 31913413
- [Derived] Golshan M, Wong SM, Loibl S, Huober JB, O'Shaughnessy J, Rugo HS, Wolmark N, Ansell P, Maag D, Sullivan DM, Metzger-Filho O, Von Minckwitz G, Geyer CE Jr, Sikov WM, Untch M. Early assessment with magnetic resonance imaging for prediction of pathologic response to neoadjuvant chemotherapy in triple-negative breast cancer: Results from the phase III BrighTNess trial. Eur J Surg Oncol. 2020 Feb;46(2):223-228. doi: 10.1016/j.ejso.2019.10.002. Epub 2019 Oct 5. PMID 31606288
- [Derived] Loibl S, O'Shaughnessy J, Untch M, Sikov WM, Rugo HS, McKee MD, Huober J, Golshan M, von Minckwitz G, Maag D, Sullivan D, Wolmark N, McIntyre K, Ponce Lorenzo JJ, Metzger Filho O, Rastogi P, Symmans WF, Liu X, Geyer CE Jr. Addition of the PARP inhibitor veliparib plus carboplatin or carboplatin alone to standard neoadjuvant chemotherapy in triple-negative breast cancer (BrighTNess): a randomised, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):497-509. doi: 10.1016/S1470-2045(18)30111-6. Epub 2018 Feb 28. PMID 29501363